CLINICAL TRIAL: NCT01279993
Title: Orthoptic Changes Following Photorefractive Keratectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Zhale Rajavi, Ophthalmic Research center
Allocation: Non-Randomized | Model: Single Group | Purpose: Supportive Care
Other Study IDs: 8659
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2008-04

CONDITIONS: Orthoptic Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kerato refractive Surgery (Experimental)
  Interventions: Procedure: Kerato refractive Surgery

INTERVENTIONS:
Procedure: Kerato refractive Surgery — This interventional case series was performed on 297 eyes of 150 patients who were candidates for PRK. Complete ophthalmic evaluations focusing on orthoptic examinations were performed before and 3 months after PRK.

SUMMARY:
Purpose: To detect orthoptic changes in patients undergoing photorefractive keratectomy (PRK). Method: This interventional case series was performed on 297 eyes of 150 patients who were candidates for PRK. Complete ophthalmic evaluations focusing on orthoptic examinations were performed before and 3 months after PRK. Results: Before PRK, two (1.3%) patients had esotropia that remained unchanged postoperatively. However, 3 (2%) patients had distance exotropia preoperatively which improved after PRK. Of 12 cases (8%) with preoperative exotropia at near, 3 (2%) cases became orthophoric. Six patients (4%) developed postoperative near exotropia. A significant reduction in means of convergence and divergence amplitudes (P<0.001) and a meaningful increase in mean of near point of convergence (NPC) (P<0.006) were noticed after PRK. A reduction of ≥10 PD in convergence amplitude and ≥5 PD in divergence amplitude were detected in 10 and 5 patients, respectively. Four patients had an preoperative NPC>10 cm which was not changed by the surgery. Out of 9 (6%) patients with baseline stereopsis >60 seconds of arc, 2 (1.33%) cases showed an improvement in stereopsis following PRK. None of the patients complained of postoperative diplopia. Conclusion: Eye deviation in patients undergoing PRK may improve or remain unchanged after operation and postoperative deviations can develop following this surgery. Diminishing of fusional amplitude and increasing of NPC as well as improving of stereopsis may also happen after PRK. Therefore, a preoperative orthoptic examination in patients with any concerning histories and/or motility issues on routine exam is recommended before performing PRK.

ELIGIBILITY:
Inclusion Criteria:

>18 yrs / refractive errors / with consent

Exclusion Criteria:

< 18 / corneal opacity - keratoconus

Dry eye / diabetes / collages vacuolar disease

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
orthoptic changes | before and after KRS
  Prism / (deviation)

SECONDARY OUTCOMES:
VA , Streopsis , deviation , fusion , NPC | before and after KRS
  Snellen , Titmus, prism, ruler

CONTACTS AND LOCATIONS:
Overall Officials: zhaleh rajavi, Assistant Professor, Principal Investigator — Imam Hossein Medical Center
Locations (1):
- Labbafinejad medical center, Tehran, Iran